CLINICAL TRIAL: NCT00680784
Title: Protocol HKT-500-US10: A Randomized, Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of HKT-500 in the Treatment of Pain Associated With Grade I or Grade II Ankle Sprain
Brief Title: HKT-500 in Adult Patients With Ankle Sprain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hisamitsu Pharmaceutical Co., Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: HKT-500-US10
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-05

CONDITIONS: Ankle Sprain
Keywords: sprain; ankle; pain
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HKT-500 Ketoprofen Topical Patch (Experimental): Randomized, double-blind, placebo-controlled, multicenter study in men and women 18 years of age or older who have a painful, acute, benign, ankle sprain of the lateral ligament(s) within the previous 48 hours.
  Interventions: Drug: HKT-500 Ketoprofen Topical Patch
- Placebo Patch (Placebo Comparator): Treatment with placebo patch
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: HKT-500 Ketoprofen Topical Patch — HKT-500 Ketoprofen Topical Patch
  Other Names: Ketoprofen Topical Patch
  Arms: HKT-500 Ketoprofen Topical Patch
Other: Placebo Patch — Placebo Patch
  Other Names: Sham treatment
  Arms: Placebo Patch

SUMMARY:
The objective of this study is to demonstrate the multiple-dose efficacy and safety of HKT-500 for the treatment of ankle sprain.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, multicenter study in men and women 18 years of age or older who have a painful, acute, benign, ankle sprain of the lateral ligament(s) within the previous 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Grade I or Grade II Ankle Sprain.

Exclusion Criteria:

* The subject is a women of childbearing potential who has a positive urine pregnancy test, who is lactating, who is not surgically sterile (by tubal ligation or hysterectomy), or at least 2 years postmenopausal, and has not practice an acceptable form of birth control (defined as the use of an intrauterine device with spermicide, a barrier method with spermicide, condoms with spermicide, subdermal implant, oral contraceptives, or abstinence) for at least 2 months prior to Visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 2 Weeks

SECONDARY OUTCOMES:
Safety Assessment | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Furuta, Study Director — Hisamitsu Pharmaceutical Co., Inc.
Locations (29):
- United States (29):
  - Hisamitsu Investigator Site., Birmingham, Alabama
  - Hisamitsu Investigator Site., Montgomery, Alabama
  - Hisamitsu Investigator Site., Anaheim, California
  - Hisamitsu Investigator Site., San Luis Obispo, California
  - Hisamitsu Investigator Site., Colorado Springs, Colorado
  - Hisamitsu Investigator Site., Kissimmee, Florida
  - Hisamitsu Investigator Site., Oldsmar, Florida
  - Hisamitsu Investigator Site., Pembroke Pines, Florida
  - Hisamitsu Investigator Site., South Miami, Florida
  - Hisamitsu Investigator Site., Blue Ridge, Georgia
  - Hisamitsu Investigator Site., Chicago, Illinois
  - Hisamitsu Investigator Site., Paducah, Kentucky
  - Hisamitsu Investigator Site., Pasadena, Maryland
  - Hisamitsu Investigator Site., Benzonia, Michigan
  - Hisamitsu Investigator Site., Cadillac, Michigan
  - Hisamitsu Investigator Site., Interlochen, Michigan
  - Hisamitsu Investigator Site., Kalamazoo, Michigan
  - Hisamitsu Investigator Site., Omaha, Nebraska
  - Hisamitsu Investigator Site., South Bound Brook, New Jersey
  - Hisamitsu Investigator Site., Albuquerque, New Mexico
  - Hisamitsu Investigator Site., New York, New York
  - Hisamitsu Investigator Site., Fargo, North Dakota
  - Hisamitsu Investigator Site., Zanesville, Ohio
  - Hisamitsu Investigator Site., Altoona, Pennsylvania
  - Hisamitsu Investigator Site., Feasterville, Pennsylvania
  - Hisamitsu Investigator Site., Morrisville, Pennsylvania
  - Hisamitsu Investigator Site., Norristown, Pennsylvania
  - Hisamitsu Investigator Site., Houston, Texas
  - Hisamitsu Investigator Site., Bellevue, Washington